CLINICAL TRIAL: NCT04159090
Title: Head- to Head Comparison of [68Ga]Ga-PSMA-11 With [18F]PSMA-1007 PET/CT in Staging Prostate Cancer Using Histopathology and Immunohistochemical Analysis as Reference-Standard
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TASMC-17-ES-0765-CTIL
Record Dates: First submitted 2019-10-29; First posted 2019-11-12 (Actual); Last update posted 2019-11-12 (Actual); Status verified 2019-11

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prostate cancer patients (Experimental)
  Interventions: Diagnostic Test: F18-PSMA

INTERVENTIONS:
Diagnostic Test: F18-PSMA — Patients with moderate or high risk of prostate cancer

SUMMARY:
PSMA (Prostate Specific Membrane Antigen) is overexpressed in prostate cancer cells.

The 68Ga-PSMA PET / CT test, using small molecules that bind to the PSMA protein and undergo intercellularization, is a test that has been shown to be more sensitive and specific than other conventional and molecular imaging modalities (CT, MRI, bone mapping, Disease in prostate cancer patients and its consequences often change therapeutic decisions in patients. In light of this, the examination of the health basket of the State of Israel was introduced to the staging of patients at moderate or high risk, as well as to the extent of the disease in patients with biochemical failure.

However, testing with 68Ga-PSMA has several limitations, resulting from the use of 68 Ga, which can be overcome by switching to fluorine-18 (18F) -based materials:

A. The generation capacity of the generator is low and therefore limits the number of tests that can be performed at a given time. In contrast, 18F is produced in cyclotron.

B. 68 Ga has a short half-life of 68 minutes, which is a logical consequence of its availability to remote medical centers from the place of production, the time of the test and the patient's comfort, and the possibility of subsequent mappings. The half-life of 18F is 110 minutes.

third. 18F has less energy than 68Ga (0.65 MEV vs. 1.9) and, as a result, a better maximum resolution that would potentially enable the demonstration of smaller lymph nodes involved in the disease.

Among the fluorine-18 (18F) materials selected for clinical application is 18F-PSMA-1007, both because the uptake is higher in the tumor than in the background, and because its removal is mainly the pathobiliary and only a small fraction of the material is released in the urine. This is another advantage of 18F-PSMA-1007 over 68Ga-PSMA, potentially enabling a better demonstration of disease sites in the pelvis, without significant absorption of the bladder material.

To date, accumulated promising experience, in Germany, in imaging with 18F-PSMA-1007. In one published case, 17 degenerative disease sites were detected in one patient with biochemical failure 9 years after undergoing radical prostatectomy, which was not demonstrated by other imaging modalities, including CT, MRI and bone mapping

ELIGIBILITY:
Inclusion Criteria:

1. Patients with prostate cancer, at moderate or high risk according to D'Amico classification during the staging phase,and who have not received any treatment (Gleason 7 and above and / or PSA> 10 and / or T2c or greater disease stage).
2. . Patients who are treated in the Department of Urology at Tel Aviv Medical Center and who are undergoing Radical Prostatectomy, as a Dependent Treatment.

Exclusion Criteria:

1. Patients with another malignant disease.
2. Patients under the age of 18 years.

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Prostate cancer can be only in males
Enrollment: 20 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2018-02-15 (Actual); Study Completion 2020-01-01 (Estimated)

PRIMARY OUTCOMES:
Patients who preformed 68Ga-PSMA-11 Biodistribution Standard to 18F-PSMA-1007 for prostate cancer. | 1 year
  The investigators will report the number of patients that preformed 68Ga-PSMA-11 Biodistribution Standard to 18F-PSMA-1007.

CONTACTS AND LOCATIONS:
Locations (1):
- Tel Aviv Sourasky medial center, Tel Aviv, Israel, Tel Aviv, Central District, Israel